CLINICAL TRIAL: NCT00337935
Title: An Open-Label, Randomized, Multi-center, Controlled Study of PROCRIT (Epoetin Alfa) for the Treatment of Anemia of Chronic Kidney Disease in the Long Term Care Setting
Brief Title: A Study of the Use of PROCRIT (Epoetin Alfa) for the Treatment of Anemia in People With Chronic Kidney Disease Who Live in Long-term Care Facilities.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Clinical Affairs, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CR012229
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Results first posted 2013-05-13 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Renal Failure , Chronic; Anemia
Keywords: Long Term Care Facilities; subcutaneous injections; PROCRIT; Epoetin alfa; Anemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — Epoetin Alfa; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epoetin Alfa (Experimental)
  Interventions: Drug: Epoetin Alfa
- Group 2 (Other): Standard treatment of anemia excluding use of erythropoetin stimulating agents (ESAs).
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: Epoetin Alfa — Epoetin alfa administered at 20,000 IU subcutaneously every 2 weeks for a period of 26 weeks
  Arms: Epoetin Alfa
Other: Standard of care
  Other Names: Standard treatment of anemia excluding use of erythropoetin stimulating agents (ESAs).
  Arms: Group 2

SUMMARY:
The purpose of this study is to show that giving PROCRIT (Epoetin alfa) every 2 weeks to increase the hemoglobin (Hb) level and then to adjust the PROCRIT (Epoetin alfa) dose every 4 weeks (Q4W) to maintain Hb levels, is safe and effective in patients with anemia from Chronic Kidney Disease (CKD), not on dialysis, who reside in long-term care facilities. In this study the frequency of PROCRIT (Epoetin alfa) dosing is under investigation.

DETAILED DESCRIPTION:
PROCRIT (Epoetin alfa) is a brand of recombinant human erythropoietin (rHuEPO). Erythropoietin is a hormone produced in the kidney. Its function is to stimulate the production of red blood cells in the bone marrow. Many patients with Chronic Kidney Disease (CKD) do not produce enough erythropoietin and thus develop anemia (a reduction in red blood cell levels). This can cause them to feel tired.

PROCRIT (Epoetin alfa) is approved by the United States Food and Drug Administration (FDA) for the treatment of anemia (low red blood cell count) in patients with CKD (not on dialysis). The approved dosing frequency for PROCRIT (Epoetin alfa) in patients with CKD is one injection three times per week. Although PROCRIT (Epoetin alfa) is approved by the FDA for the treatment of certain types of anemia at different dosing schedules, the dosing schedules that will be used in this study are investigational in CKD. An investigational use is one that is currently not approved by the FDA.

This is an open-label, randomized (patients are assigned different treatments based on chance), multi-center, controlled study of patients with anemia of Chronic Kidney Disease (CKD), not on dialysis, who reside in long-term care facilities. Approximately 156 patients with CKD, not on dialysis, who have not received an erythropoietin receptor agonist (a drug that stimulates red blood cell production) for eight weeks immediately prior to screening (Week -1) and who have a hemoglobin (Hb, a measure of the number of red blood cells), less than 11 g/dL at screening will be eligible to participate. Patients will be evaluated for eligibility during a one-week screening phase. Eligible patients will be randomized in a 3:1 ratio to a PROCRIT (Epoetin alfa) group or to the control group for a period of 26 weeks. Randomization is done through a computer that randomly assigns the subject by chance (like rolling dice) to one of two groups (No one can choose the group to which they will be assigned.). They will have a 3 to 1 chance of being assigned to Group 1 versus Group 2, which means that out of every 4 patients entering the study 3 will receive PROCRIT (Epoetin alfa) and 1 will not.

Group 1 -will receive PROCRIT (Epoetin alfa) 20,000 Units (U) every 2 weeks until the hemoglobin reaches 11.0 g/dL or higher and remains at this level for two measurements in a row. At Week 6 or thereafter, the 20,000 Unit dose may be adjusted upward or downward as required to obtain the two consecutive hemoglobin measurements. Once the two consecutive measurements have been achieved, PROCRIT (Epoetin alfa) will be given every 4 weeks (Q4W) at double the previous dose to obtain a target hemoglobin of up to 12.0 g/dL. There will be no conversion to Q4W before Week 6 or after Week 18. If the hemoglobin drops, patients may go back to receiving PROCRIT (Epoetin alfa) every 2-weeks. If the hemoglobin rises above 12.0 g/dL, patients will not receive another dose of PROCRIT (Epoetin alfa) until the Hg level is below 12.0 g/dL. If the hemoglobin rises rapidly, patients will not receive another dose of PROCRIT (Epoetin alfa) until the rise is 1 g/dL or less in a 2-week period. The maximum amount of PROCRIT (Epoetin alfa) that this group can receive is 60,000 Units over a 4-week period. All doses of PROCRIT (Epoetin alfa) are injected under the skin (subcutaneous).

Group 2 - will not receive any PROCRIT (Epoetin alfa). This group will continue to receive the care that they are now receiving from their physician and the physician will review all lab results.

Since a lack of iron could interfere with the ability of patients to make red blood cells, patients in both groups will have iron levels checked at the screening visit and during the study. Based on the results of iron tests, the study doctor may prescribe an oral (by mouth) or intravenous (injection) iron supplement during the study. If the need for iron supplementation is determined, patients will receive iron supplementation no matter which group they are in.

Every two weeks a study visit will be performed. At each visit, blood pressure and heart rate will be checked, and blood will be drawn for all patients and sent to the central laboratory for complete blood count (CBC). The Hb by CBC will be used for efficacy analysis ( to measure the effectiveness of the study drug in increasing the hemoglobin level). Hb testing by HemoCue will be performed every two weeks on-site for PROCRIT (Epoetin alfa) group patients, for the purpose of real-time dosing decisions. (HemoCue is the brand name of a portable hemoglobin test that uses a drop of blood to obtain immediate hemoglobin measurements). PROCRIT (Epoetin alfa) will be administered at a dose based on the HemoCue Hb measurement. Full hematology panel, serum chemistry, and iron status will be assessed at intervals throughout the study by a central laboratory. The number of units of packed red blood cells (PRBC) transfused, pre-transfusion Hb level, and the reasons for transfusion will be collected. Hemoglobin response will also be measured. A patient exhibiting a hemoglobin response will have two consecutive Hb measurements at least 1 g/dL greater than baseline any time during the study or have two consecutive Hb measurements >= 11.0 g/dL at any time during the study. Falls, activities of daily living (ADLs), and mobility will be assessed during the study. Clinical laboratory results, blood pressure and heart rate, and the incidence and severity of adverse events will be monitored during the study.

The study hypothesis is that the mean Hb change from baseline to the end of study will be significantly higher in the PROCRIT (Epoetin alfa) group over the control group. Group 1 patients will receive a maximum of 13 doses of PROCRIT (Epoetin alfa) by subcutaneous injection (under the skin) for up to 26 weeks. Dosage is based on the hemoglobin measurement done at each visit. Doses will be started at an every 2-week interval and may be increased to every four weeks. The maximum dose that can be given is 60,000 Units of PROCRIT (Epoetin alfa) over a 4-week period. Any PROCRIT (Epoetin alfa) dose over 40,000 Units will be administered in two separate injections.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Kidney Disease (CKD) Stage 3, 4, or 5 (not on dialysis), Glomerular Filtration Rate (GFR) [<60 mL/min/1.73 m2], or CKD Stage 2 (GFR 61-90 mL/min/1.73 mm2) with evidence of kidney damage (defined as structural or functional abnormalities of the kidneys) for greater than 3 months
* Hb <11 g/dL measured at screening and a stable creatinine over the last 3 months
* expected to stay in a Long Term Care (LTC) facility for at least six months
* not receiving erythropoietic agents within eight weeks prior to screening.

Exclusion Criteria:

* No significant hematological disease (including, but not limited to, myelodysplastic syndrome, hematological malignancy, hemolytic syndromes, hemoglobinopathy), or with a current diagnosis of anemia due to blood loss (e.g., hemolysis or gastrointestinal bleeding) or any cause of anemia other than CKD (e.g., hypothyroidism, HIV)
* No history of deep venous thrombosis (DVT) or pulmonary embolus (PE) within 12 months prior to screening (prior superficial thrombophlebitis is not an exclusion criterion), or a history of cerebrovascular accident (CVA), transient ischemic attack (TIA), Acute Coronary Syndrome (ACS), or other arterial thrombosis within 6 months before study entry. [ACS includes Unstable Angina, Q wave Myocardial Infarction and non-Q wave Myocardial Infarction]
* No uncontrolled or severe cardiovascular disease including uncontrolled hypertension (systolic BP > 170 mm/Hg, or diastolic BP > 100 mm/Hg), or congestive heart failure (New York Heart Association (NYHA) Class IV)
* No known solid tumor malignancy, receiving chemotherapy for cancer or having major surgery within one month prior to screening or expected during study participation
* No history of receiving a transplanted organ, or scheduled to receive an organ transplant during the course of the study, with the exception of a corneal transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2006-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Standard treatment of anemia excluding use of erythropoietin stimulating agents (ESAs).
- PROCRIT (Epoetin Alfa): epoetin alfa administered at 20,000 IU subcutaneously every 2 weeks for a period of 26 weeks
Period: Overall Study
Arm/Group | Standard of Care | PROCRIT (Epoetin Alfa)
Started | 39 | 118
Completed | 29 | 91
Not Completed | 10 | 27
Not completed — Adverse Event | 2 | 5
Not completed — Death | 2 | 8
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 4 | 3
Not completed — Withdrawal by Subject | 1 | 7
Not completed — Other | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | PROCRIT (Epoetin Alfa) | Total
Number analyzed (Participants) | 39 | 118 | 157
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 6
  >=65 years | 37 | 114 | 151
Age Continuous [Mean (Standard Deviation); unit: Years] | 84.4 (10.9) | 84.1 (9.2) | 84.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 90 | 123
  Male | 6 | 28 | 34

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hemoglobin Level From Baseline to the End of Study (26 Weeks)
Time Frame: Week 0 to Week 26
Population: Modified intent to treat (mITT) - all subjects with at least 1 hemoglobin measurement after baseline. Four subjects did not have hemoglobin measurement post baseline.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Standard of Care | PROCRIT (Epoetin Alfa)
Number analyzed (Participants) | 39 | 114
g/dL | 0.3 (1.3) | 0.9 (1.0)
Statistical Analysis 1: Comparison: Standard of Care vs PROCRIT (Epoetin Alfa); Test type: Superiority or Other; p = .0062, ANCOVA — a priori theshold for statistical significance was p=0.05; Baseline Hemoglobin was used as a covariate; Mean Difference (Net) = 0.6, 95% CI 2-sided [0.2 to 0.9], Standard Error of Mean .2

2. Secondary Outcome: The Number of Patients Achieved a Hemoglobin Response.
Description: Hemoglobin reponse was defined as 2 consecutive hemoglobin measurements at least 1.0 g/dL above baseline or 2 consecutive hemoglobin measurements at least 11.0 g/dL
Time Frame: Week 0 to Week 26
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Standard of Care | PROCRIT (Epoetin Alfa)
Number analyzed (Participants) | 39 | 114
participants | 21 | 97
Statistical Analysis 1: Comparison: Standard of Care vs PROCRIT (Epoetin Alfa); Test type: Superiority or Other; p < 0.001, Chi-squared — A priori threshold for statistical significance p=0.05

3. Secondary Outcome: Time to Hemoglobin Response
Description: Time to hemoglobin reponse was defined as the time between individual treatment start date and the first of 2 consecutive hemoglobin measurements at least 1.0 g/dL above baseline or 2 consecutive hemoglobin measurements at least 11.0 g/dL. Note: Upper 95% confidence limit for the Standard of Care Group was not estimable because an insufficient number of participates reached the event at the final time point for assessment.
Time Frame: Week 0 to Week 26
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Standard of Care: Standard treatment of anemia excluding use of erythropoietin stimulating agents (ESAs). Upper 95% confidence limit for the Standard of Care Group was not estimable because an insufficient number of participates reached the event at the final time point for assessment.
Arm/Group | Standard of Care | PROCRIT (Epoetin Alfa)
Number analyzed (Participants) | 39 | 114
Days | 114 [43 to NA] — Upper 95% confidence limit for the Standard of Care Group was not estimable because an insufficient number of participates reached the event at the final time point for assessment. | 41 [29 to 43]
Statistical Analysis 1: Comparison: Standard of Care vs PROCRIT (Epoetin Alfa); Test type: Superiority or Other; p < 0.0001, Log Rank — A priori threshold for statistical significance p=0.05

ADVERSE EVENTS:
Time Frame: 26 weeks or early withdraw
Description: Any ongoing adverse events were followed up to 30 days and serious adverse events until resolution. Serious adverse events were to be reported throughout the study including those serious adverse events spontaneously reported within 30 days after the patient completed the study.
Arm/Group | Standard of Care | PROCRIT (Epoetin Alfa)
Serious Adverse Events (participants affected / at risk) | 14/39 | 39/118
Other Adverse Events (participants affected / at risk) | 34/39 | 99/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=39) | PROCRIT (Epoetin Alfa) (N=118)
Acute Myocardial Infarction (Cardiac disorders) | 3 | 1
Atrrial Fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 2 | 4
Cardiopulmonary Failure (Cardiac disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Joint Abscess (Infections and infestations) | 0 | 1
Oesteomyelitis (Infections and infestations) | 1 | 0
Pneumococcal Bacteraemia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 5
Pneumonia Pneumococcal (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 1
Staphylococcal Sepsis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 4
Wound Infection Staphylococcal (Infections and infestations) | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 2
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 1
Therapeutic Agent Toxicity (Injury, poisoning and procedural complications) | 1 | 0
Anticonvulsant Drug Level Decreased (Investigations) | 0 | 1
Haemoglobin Decreased (Investigations) | 0 | 1
International Normalised Ratio Increased (Investigations) | 1 | 0
Weight Decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Failure To Thrive (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dementia (Nervous system disorders) | 1 | 2
Dementia Alzheimer's Type (Nervous system disorders) | 1 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Transient Ischaemic Attack (Nervous system disorders) | 0 | 2
Aggression (Psychiatric disorders) | 1 | 1
Renal Failure (Renal and urinary disorders) | 3 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 5
Renal Failure Chronic (Renal and urinary disorders) | 1 | 0
Urethral Perforation (Renal and urinary disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic Embolus (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Urosepsis (Infections and infestations) | 2 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=39) | PROCRIT (Epoetin Alfa) (N=118)
Conjunctivitis (Eye disorders) | 2 | 4
Abdominal Pain (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 4 | 6
Diarrhoea (Gastrointestinal disorders) | 6 | 19
Dysphagia (Gastrointestinal disorders) | 2 | 7
Nausea (Gastrointestinal disorders) | 2 | 10
Vomiting (Gastrointestinal disorders) | 8 | 22
Localised Oedema (General disorders) | 2 | 0
Oedema Peripheral (General disorders) | 5 | 13
Bronchitis (Infections and infestations) | 0 | 6
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 20
Urinary Tract Infection (Infections and infestations) | 9 | 21
Contusion (Injury, poisoning and procedural complications) | 6 | 17
Excoriation (Injury, poisoning and procedural complications) | 4 | 8
Open Wound (Injury, poisoning and procedural complications) | 2 | 5
Skin Laceration (Injury, poisoning and procedural complications) | 6 | 24
Dehydration (Metabolism and nutrition disorders) | 4 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 11
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 | 12
Lethargy (Nervous system disorders) | 2 | 5
Insomnia (Psychiatric disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 8
Blister (Skin and subcutaneous tissue disorders) | 2 | 7
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 3 | 5
Erythema (Skin and subcutaneous tissue disorders) | 4 | 5
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 9
Rash (Skin and subcutaneous tissue disorders) | 2 | 11
Scab (Skin and subcutaneous tissue disorders) | 2 | 1
Skin Irritation (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 0 | 7
Hypotension (Vascular disorders) | 2 | 5
Weight Decreased (Investigations) | 4 | 9

LIMITATIONS AND CAVEATS:
Upper 95% confidence limit for the Standard of Care Group was not estimable because an insufficient number of participates reached the event at the final time point for assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes